CLINICAL TRIAL: NCT00936507
Title: Does Portion Size Influence Intake of Low-Energy-Dense Foods in Preschool-aged Children?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1-Smith
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Caloric Intake
Keywords: energy density; portion size; child feeding
MeSH Terms: interventions — Portion Size

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Low-ED, small portion (Experimental)
  Interventions: Other: Energy Density/Portion Size
- Low-ED, large portion (Experimental)
  Interventions: Other: Energy Density/Portion Size
- High-ED, small portion (Experimental)
  Interventions: Other: Energy Density/Portion Size
- High-ED, large portion (Experimental)
  Interventions: Other: Energy Density/Portion Size

INTERVENTIONS:
Other: Energy Density/Portion Size

SUMMARY:
The purpose of this randomized controlled study using a crossover design is to investigate the main effect of portion size and food type (low-energy dense vs. high-energy dense) on caloric intake.

DETAILED DESCRIPTION:
The purpose of this investigation is to examine the impact of portion size on intake of a low energy dense food (fruit). Preschool-aged children will be provided with a small and large portion of applesauce (low-energy-dense food) and chocolate pudding (higher-energy-dense food) and allowed to eat the foods ad libitum during an afternoon snack in their usual preschool classroom. Measures of the amount of each food (grams and kilocalories) consumed will be taken.

The following hypotheses are proposed:

1. A significant main effect of portion size will occur, such that children will consume more food, both in grams and kilocalories, in the large portion as compared to the small portion conditions.
2. A main effect of food type on caloric intake will occur, such that children will consume less calories in the applesauce condition as compared to the pudding condition, due to the differences in energy density of these foods. It is not anticipated that a difference in grams consumed from each food will occur.

ELIGIBILITY:
Inclusion Criteria:

* All children that are ≥3 years of age enrolled in the ELC preschool with parental consent can participate.
* Eligible children must also like both the applesauce and the pudding, and be able to consume foods with a spoon.

Exclusion Criteria:

* Children allergic to applesauce or chocolate pudding or who are lactose- intolerant will not be included in the study.
* Did not attend all feeding sessions.
* Did not consume more than 5 grams from any of the foods on an occasion.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Healthy Eating and Activity Laboratory, University of Tennessee, Knoxville, Tennessee, United States